CLINICAL TRIAL: NCT05972473
Title: A Phase 3, Randomized, Double-masked, Active-Controlled Study to Evaluate the Efficacy and Safety of Intravitreal IBI302(Efdamrofusp Alfa) in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: A Study to Evaluate the Efficacy and Safety of IBI302 in Subjects With nAMD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI302A301CN
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — IBI302

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept (Active Comparator): Drug: Aflibercept 2mg/eye; Intraocular injection
  Interventions: Drug: Aflibercept Ophthalmic
- IBI302 dose 8mg (Experimental): Drug: IBI302 8mg/eye; Intraocular injection
  Interventions: Biological: IBI302

INTERVENTIONS:
Drug: Aflibercept Ophthalmic — 2mg Aflibercept will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive monthes, folloesd by once every 8 weeks(Q8W).
  Arms: Aflibercept
Biological: IBI302 — 8 mg IBI302 will be administered by intraitreal injection into the study eye at intervals as specified in the study protocol.
  Arms: IBI302 dose 8mg

SUMMARY:
The study is designed for multi-center,randomized,double-masked,active-contralled study to evaluate effective and security of intravitreal injection of IBI302 in subjects with neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to study participation;
2. Male or female ≥ 50 years of age at the time of signing the informed consent;
3. Active subfoveal CNV secondary to nAMD, or active CNV with intra/subretinal fluid involving the fovea;
4. BCVA of 19 to 78 ETDRS letters (inclusive) in the study eye at baseline.

Exclusion Criteria:

1. Ocular disease:

   * Any concurrent intraocular condition/systemic disease in the study eye at screening or baseline that, in the judgment of the investigator, may cause the participant fail to respond to the treatment or confuse the interpretation of study results;
   * Total lesion area(including blood, atrophy, fibrosis, PED and neovascularization)> 12 optic disc area (DA) on FFA;
   * Subretinal hemorrhage area > 50% of the total lesion area, or subretinal hemorrhage area involving macular fovea ≥ 1 DA;
   * Fibrosis or atrophy area > 50% of the total lesion area, or involving the fovea; Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg after standard treatment);
   * Presence of active intraocular or periocular infection or inflammation;
2. Ocular treatment:

   * Anti-VEGF or anti-complement therapy in the study eye within 90 days prior to baseline;
   * Fundus laser photo-coagulation in the study eye within 90 days prior to baseline;
   * Photodynamic Therapy (PDT) in the study eye within 90 days prior to baseline;
   * History of vitreoretinal surgery, penetrating keratoplasty in the study eye;
3. General condition or treatment:

   * Uncontrolled hypertension (defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg after standard treatment);
   * HbA1c > 8% within 28 days prior to baseline; Systemic anti-VEGF drug and anti-complement drug therapy within 90 days prior to baseline;
   * History of hypersensitivity to any component of the test article, control article, or clinically relevant sensitivity to fluorescein dye, povidone-iodine;
   * Pregnant or lactating women; Inappropriate for the study (e.g., substance abuse, inability or unwillingness to follow the trial protocol), as judged by the investig.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Best corrected visual acuity ( BCVA ) in the study eye. | At week 44, 48, 52
  Change from Baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) letter score at week 44, 48, 52.

SECONDARY OUTCOMES:
The proportion of participants with absence intraretinal fluid (IRF) and absence subretinal fluid (SRF) in the fovea at Week 16 | At week 16
  The intraretinal fluid and subretinal fluid is measured by optical coherence tomography (OCT) in the central subfield(center 1 millimeter)
Change from baseline in BCVA at Week 52 and 100 | Upto Week 100
  Best corrected visual acuity (BCVA) was measured on early treatment diabetic retinopathy study(ETDRS) chart at a starting distance of 4 meters. The BCVAletter score ranges from 0 to 100(best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Change from baseline in central subfield thickness (CST) measured by optical coherence tomography (OCT) at Week 52 and 100 | Upto Week 100
  Central subfield thickness was defined as the distance between the internal limiting member and the Bruch's member using OCT, as assessed by the central reading center.
Change from baseline in area of CNV on fundus fluorescence angiography (FFA) at Week 52 and 100 | Upto Week 100
  the area of the choroidal neovascularization lesion in the study eye was measured by a central reading center using FFA
Proportion of participants on a q8W, q12W, and q16W treatment intervals at Week 52 and 100 | Upto Week 100
  Percentages are based on number of participants randomized to the IBI302 group who have not discontinued the study at week 52 and 100. the treatment interval at a givven visit is defined as the treatment interval decision followed at that visit.
Incidence, relatedness to the study drug and severity of ocular and Non-ocular adverse events (AE), treatment emergent adverse events (TEAE) and serious adverse events (SAE). | Upto Week 100
  All AEs were recorded and the investigator made an assessment of seriousness,severity, and causality of each AE.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No